CLINICAL TRIAL: NCT04404218
Title: Randomized Clinical Trial of Açaí Palm Berry Extract as an Intervention in Patients Diagnosed With COVID-19
Brief Title: The Açaí Berry COVID-19 Anti-Inflammation Trial
Acronym: ACAI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Michael Farkouh, Chair & Director, Peter Munk Centre of Excellence in Multinational Clinical Trials, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTO3176
Record Dates: First submitted 2020-05-24; First posted 2020-05-27 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: COVID
Keywords: açaí berry; COVID; community care patients

STUDY DESIGN:
Intervention Model Description: Prospective, double-blinded, placebo-controlled, randomized, multicentre clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinding, using placebo pills.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Açaí palm berry extract (Experimental): Açaí palm berry extract is a powerful antioxidant with no known side-effects and is widely consumed in Brazil. Açaí palm berry chemical composition has been established and includes several antioxidants - gallic acid, catechin, chlorogenic acid, caffeic acid, p-coumaric acid, epicatechin, orientin, cyanidin-3-0-glucoside, luteolin and apigenin. Orientin is the most concentrated compound (7,96mg/g) and this compound is able to modulate the NLRP3 inflammasome.
  Interventions: Dietary Supplement: Açaí palm berry extract - natural product
- Placebo arm (Placebo Comparator): This study will be double-blinded and placebo-controlled. To ensure double-blinding, placebo and active compound capsules will be over-encapsulated with DBCAPS® capsules, which were developed with a tamper-evident design to address the clinical trial challenges of testing without bias. These capsules are made of gelatin and have no interaction with bioavailability.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Açaí palm berry extract - natural product — Patients will be prescribed to take 1 capsule (520mg) of Açaí Palm Berry every 8 hours for a total of 3 capsules a day, during 30 days. Total dose: 1,560mg/day of Açaí Berry extract.
  Arms: Açaí palm berry extract
Other: Placebo — Patients will take 1 placebo pill every 8 hours (total of 3 capsules a day) for 30 days.
  Arms: Placebo arm

SUMMARY:
The Açaí trial will be testing if the açaí berry extract, a safe natural product with anti-inflammatory properties, can be used as a treatment option in adult patients with COVID-19 in the community.

DETAILED DESCRIPTION:
The current COVID-19 pandemic is caused by the novel coronavirus (SARS-Cov-2). The virus origins have been studied and evidence so far suggests it originates in bats, with spread to humans likely mediated by an intermediate mammalian. Bats have a dampened Nod-like receptor family, pyrin-containing 3 (NLRP3)-mediated inflammation. Dampening NLRP3-mediated inflammation has been associated with the asymptotic viral status, therefore it is plausible that the pathogenic inflammatory response of SARS-CoV-2 might be associated with activation of NLRP3 inflammasome. Data show that the natural extract of Açaí Palm Berry (Euterpe oleracea Mart.) is a potent inhibitor of NLRP3. This is a safe, inexpensive, and readily available natural health supplement which could be a rapid response treatment intervention for patients with COVID-19.

Our primary objective is to establish whether açai palm berry extract (Euterpe oleracea), given to community-dwelling adult patients diagnosed with COVID-19, compared to placebo, improves outcomes over 30 days on the 7-point ordinal scale described by Cao et al, and which is being used widely in COVID-19 trials with the aim of harmonizing endpoints. This study will be a prospective, double-blinded, placebo-controlled, randomized, multicentre clinical trial of Açaí Palm Berry extract in adult patients tested positive for SARS-Cov-2 in the last 7 days and that are currently being treated in the outpatient setting. The intervention group will receive 3 capsules of 520mg (one capsule every eight hours) of Acai Palm Berry extract (Nature's Way, NPN80038874) for 30 days. The non-intervention group will receive placebo pills, on top of standard clinical care. Our main endpoint will be the 7-point ordinal scale.

This project has the benefit of offering a safe and widely used natural extract as a potential treatment strategy to decrease inflammation and improve disease outcomes in patients with COVID-19. With no vaccine currently available, the search for effective treatments is a timely approach. The potential impact of such a therapeutic agent, if effective, can be quite vast given that it can be readily used by anyone and, most importantly, is affordable in many countries.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 40 years of age; and
* Mild to moderate symptoms including fever, dry cough, and tiredness; and
* Tested positive for SARS-Cov-2, via virological diagnosis (PCR), in the last 7 days; and
* Not hospitalized at the time of randomization, with no limitations on activities; and
* Willingness to complete questionnaires and records associated with the study.

Exclusion Criteria:

* Hospitalized patients at the time of enrollment; or
* Known allergy to study medication or its non-medicinal ingredients; or
* Currently taking açai extract or juice; or
* Chronic severe renal impairment (creatinine clearance <30 mL/min or on renal replacement therapy); or
* Pregnant or breastfeeding patients; or
* Women who are planning to become pregnant during the study; or
* End-stage cancer or patients in whom imminent demise is anticipated and there is no commitment to active ongoing intervention; or
* Unable to provide informed consent; or
* Patients taking antiplatelet/blood-thinning medication; or
* Patients with unstable metabolic disease/chronic diseases/ diseases with any comorbidities and/or any serious medical condition or abnormality of clinical laboratory tests that precludes the patient's safe participation in and completion of the study or puts them in a greater risk of developing severe symptoms (e.g. Individuals with an acute infectious disease, immune-compromised, self-reported confirmation of HIV, other lung diseases such as asthma, emphysema, neurological conditions); or
* Patients who participated in other clinical research studies 30 days prior to screening; or
* Patients who are participating in another clinical trial at the same time.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2020-08-04 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
7-point ordinal symptom scale | 30 days
  Symptom comparison between patients from the treatment vs control group, using an ordinal symptom scale based on the WHO scale. Patients who were hospitalized will be classified according to their worst score over 30 days and non-hospitalized patients according to their score at 30 days.

SECONDARY OUTCOMES:
The composite of all-cause mortality and need for mechanical ventilation | 30 days
  First occurrence of all-cause mortality or need for mechanical ventilation
The composite of all-cause mortality and hospitalization | 30 days
  First occurrence of all-cause mortality or hospitalization
All-cause mortality | 30 days
  All-cause mortality
Need for mechanical ventilation | 30 days
  Need for mechanical ventilation
Need for hospitalization | 30 days
  Need for hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Michael Farkouh, MD, MSc, Principal Investigator — Peter Munk Cardiac Centre; University Health Network; University of Toronto; Ana Andreazza, PhD, Principal Investigator — Department of Pharmacology & Toxicology; University of Toronto
Locations (3):
- Brazil (2):
  - Instituto de Pesquisas em Saude (IPS)/ Universidade de Caxias do Sul (UCS), Caxias do Sul, Rio Grande do Sul
  - Instituto Prevent Senior (IPS) - Hospital Sancta Maggiore, São Paulo, São Paulo
- Heart Health Institute Research Inc, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Machado AK, Andreazza AC, da Silva TM, Boligon AA, do Nascimento V, Scola G, Duong A, Cadona FC, Ribeiro EE, da Cruz IB. Neuroprotective Effects of Acai (Euterpe oleracea Mart.) against Rotenone In Vitro Exposure. Oxid Med Cell Longev. 2016;2016:8940850. doi: 10.1155/2016/8940850. Epub 2016 Oct 3. PMID 27781077
- [Background] Machado AK, Cadoná FC, Assmann CE, Andreazza AC, Duarte MMMF, Branco CS, Zhou X, Souza DV, Ribeiro EE, Cruz IBM. Açaí (Euterpe oleracea Mart.) has anti-inflammatory potential through NLRP3-inflammasome modulation. Journal of Functional Foods. Volume 56, 2019, Pages 364-371, https://doi.org/10.1016/j.jff.2019.03.034.
- [Background] Kim HK, Chen W, Andreazza AC. The Potential Role of the NLRP3 Inflammasome as a Link between Mitochondrial Complex I Dysfunction and Inflammation in Bipolar Disorder. Neural Plast. 2015;2015:408136. doi: 10.1155/2015/408136. Epub 2015 May 13. PMID 26075098
- [Background] Kim HK, Andreazza AC, Elmi N, Chen W, Young LT. Nod-like receptor pyrin containing 3 (NLRP3) in the post-mortem frontal cortex from patients with bipolar disorder: A potential mediator between mitochondria and immune-activation. J Psychiatr Res. 2016 Jan;72:43-50. doi: 10.1016/j.jpsychires.2015.10.015. Epub 2015 Oct 26. PMID 26540403
- [Background] Ulbricht C, Brigham A, Burke D, Costa D, Giese N, Iovin R, Grimes Serrano JM, Tanguay-Colucci S, Weissner W, Windsor R. An evidence-based systematic review of acai (Euterpe oleracea) by the Natural Standard Research Collaboration. J Diet Suppl. 2012 Jun;9(2):128-47. doi: 10.3109/19390211.2012.686347. PMID 22607647
- [Background] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464